CLINICAL TRIAL: NCT04831138
Title: A Prospective Study to Evaluate Quantitative Non-Contrast Perfusion Using Arterial Spin Labeled MR Imaging for Assessment of Therapy Response in Metastatic Renal Cell Carcinoma
Brief Title: Non-Contrast Perfusion Using Arterial Spin Labeled MR Imaging for Assessment of Therapy Response in Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The treatment landscape changed and hence unable to recruit patients undergoing only anti-angiogenic treatment.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ananth Madhuranthakam, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 032018-078; 1U01CA207091-01A1 (NIH)
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma
Keywords: magnetic resonance imaging; arterial spin labeling
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCC Patients (Experimental): Patients with locally advanced or metastatic renal cell carcinoma
  Interventions: Other: MRI with ASL
- Healthy Volunteers (Other): Healthy volunteers to optimize protocol
  Interventions: Other: ASL-MRI

INTERVENTIONS:
Other: MRI with ASL — T0 (Week 0): MRI with ASL will be performed either for research alone or along with patient's standard of care imaging session including contrast-enhancement.
  T1 (Day 7+-2): contrast-enhanced research MRI with ASL T2 (Day 14+-2): contrast-enhanced research MRI with ASL T3: MRI with ASL will be performed along with patient's standard of care imaging session.
  T4: MRI with ASL will be performed along with patient's standard of care imaging session.
  T5: MRI with ASL will be performed along with patient's standard of care imaging session.
  Other Names: MR Imaging
  Arms: RCC Patients
Other: ASL-MRI — Healthy volunteers - MRI with ASL protocol optimization
  Other Names: MRI Optimization
  Arms: Healthy Volunteers

SUMMARY:
Magnetic Resonance Imaging (MRI) including Arterial Spin Labeling (ASL) will be performed before, during, and after the treatment, in a total of up to 6 MRI sessions until 7 months after the first session, or when progression is clinically indicated. Thereafter, patients will be followed through standard clinical examinations for the next 3 years or until demise, whichever occurs first.

Clinically, metastatic renal cell carcinoma (RCC) patients are imaged every 2-3 months after the initiation of anti-angiogenic therapy, since morphological (i.e. size) changes are not anticipated earlier. However, our preliminary experience has shown functional changes including perfusion as early as 2-weeks after the initiation of the treatment. T0, T1, and T2 sessions will be performed for this proposal, while T3, T4, and T5 will be performed along with the clinical imaging sessions. All MR imaging sessions will be scheduled within ±1 or ±2 weeks of the target time period.

The research MR imaging may take approximately an additional 15 minutes per each imaging session, when done in conjunction with the clinical imaging. The T0, T1, and T2 research MR imaging sessions will be performed additionally for the purpose of this study, with each taking approximately one hour.

DETAILED DESCRIPTION:
The incidence of kidney cancer has steadily increased over the past three to four decades and is among the 10 most frequently diagnosed cancers in the US. Approximately 63,990 new cases of kidney cancer are estimated in 2017 and the prognosis has been historically poor. The current 5-year survival rates are estimated at 74% overall, decreasing to 53% among patients with locally advanced diseases.

The most common form of kidney cancer, renal cell carcinoma (RCC), occurs in 90% of all kidney cancers. Among patients with localized RCC who are treated with nephrectomy, approximately one quarter have relapses in distant sites. Among patients with metastatic RCC, the 5-year survival rates are approximately 8%. With better understanding of the pathogenesis of the most common type of RCC, clear-cell renal cell carcinoma (ccRCC), newer treatment options with new agents are being developed to increase survival rates.

The high cost and potential risks associated with human trials for the newly developed experimental therapies have emphasized the need for sensitive monitoring of tumor response. Imaging approaches can play an important role in the evaluation and selection of potential new therapies with non-invasive longitudinal monitoring of treatment response. Currently, the radiological assessment of treatment outcomes predominantly relies on morphological (i.e. size) changes using the Response Evaluation Criteria in Solid Tumors (RECIST) and other similar scores. This is a major limiting factor as the effects of many therapeutic agents at the microscopic level precede the eventual changes in tumor size. One such tumor property that has gained increased attention is angiogenesis, which has been shown to support tumor proliferation and infiltration. Increasing numbers of clinical trials have begun targeting tumor vascular supplies by directly inhibiting angiogenesis (e.g. antiangiogenic therapy). Such clinical trials and the eventual clinical use of these therapies would be greatly assisted by the availability of robust imaging indicators of angiogenesis (i.e. tissue perfusion).

Positron Emission Tomography (PET) using 15O-labeled water (15O-PET) is considered the gold standard for non-invasive measurement of tissue perfusion. However, the use of 15O-PET requires a cyclotron in close proximity to PET to produce short lived 15O-water (half life 2.4 min), limiting its applicability in clinical settings. Alternative imaging techniques include ultrasound using microbubbles, perfusion computed tomography (CT) using iodinated contrast agent and perfusion MRI using gadolinium based contrast agents. All of these techniques require exogenous agents, restricting their use in longitudinal monitoring of treatment response.

ASL-MRI has recently emerged as a quantitative imaging (QI) method to measure perfusion (or capillary blood flow) without the administration of exogenous contrast agents. ASL magnetically "labels" the highly permeable water in the blood as a tracer and measures their accumulation in the tissue of interest, without injecting any exogeneous contrast. Various versions of ASL have been validated in animals using microspheres, and in humans using 15O-PET in the brain. ASL also has a number of advantages compared to dynamic contrast enhanced (DCE) and dynamic susceptibility contrast (DSC) based MR perfusion measurements. Specifically, ASL does not require exogenous agent alleviating the concerns of gadolinium accumulation or nephrogenic systemic fibrosis (NSF) in patients with impaired renal function and, unlike DCE/DSC, the contribution of vascular permeability to ASL measured perfusion is negligible enabling absolute perfusion quantification in physiological units.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic renal cell carcinoma.
* Patients scheduled to undergo anti-angiogenic treatment or immunotherapy
* Eastern Cooperative Oncology Group (ECOG) Status 0, 1 and 2.
* Women of child-bearing potential must agree to undergo a urine pregnancy screening per standard Radiology departmental protocol, in place to prevent imaging of pregnant patients. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: 1) Has not undergone a hysterectomy or bilateral oophorectomy; or 2) Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects may not be receiving any other anti-angiogenic agents, at the time of enrollment.
* Subjects must not be pregnant since pregnancy is a contraindication to administration of gadolinium-based contrast agents.
* Any contraindication to MRI per Radiology Department's routine protocol, e.g. MRI-incompatible objects, including but not limited to medical devices (e.g. pacemakers, automated implantable cardioverter defibrillators, etc.) and other foreign bodies.
* Known severe allergic reaction to Gadolinium-based contrast agents.
* Patients with sickle cell disease and patients with other hemolytic anemias (low red blood count in body).
* Patients with uncontrollable claustrophobia, severe lower back pain, and uncontrollable tremors, to the point that it would render them unable to tolerate an MRI study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Renal Cell Carcinoma (RCC) Patients: Patients with locally advanced or metastatic renal cell carcinoma
  Magnetic Resonance Imaging (MRI) with Arterial Spin Labeling (ASL): T0 (Week 0): MRI with ASL will be performed either for research alone or along with patient's standard of care imaging session including contrast-enhancement.
  T1 (Day 7+-2): contrast-enhanced research MRI with ASL T2 (Day 14+-2): contrast-enhanced research MRI with ASL T3: MRI with ASL will be performed along with patient's standard of care imaging session.
  T4: MRI with ASL will be performed along with patient's standard of care imaging session.
  T5: MRI with ASL will be performed along with patient's standard of care imaging session.
Period: Overall Study
Arm/Group | Renal Cell Carcinoma (RCC) Patients | Healthy Volunteers
Started | 2 | 4
Completed | 0 | 4
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- RCC Patients: Patients with locally advanced or metastatic renal cell carcinoma
  MRI with ASL: T0 (Week 0): MRI with ASL will be performed either for research alone or along with patient's standard of care imaging session including contrast-enhancement.
  T1 (Day 7+-2): contrast-enhanced research MRI with ASL T2 (Day 14+-2): contrast-enhanced research MRI with ASL T3: MRI with ASL will be performed along with patient's standard of care imaging session.
  T4: MRI with ASL will be performed along with patient's standard of care imaging session.
  T5: MRI with ASL will be performed along with patient's standard of care imaging session.
- Total: Total of all reporting groups
Arm/Group | RCC Patients | Healthy Volunteers | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Perfusion in the Tumor
Description: Measure change in perfusion at 7 days and 14 days compared to baseline measurement.
Time Frame: Baseline to 7 and 14 days
Population: Data were not collected and analyzed due to termination of the study and the 2 RCC patients enrolled not completing the study.
Groups:
- RCC Patients: Patients with locally advanced or metastatic renal cell carcinoma
  MRI with ASL: T0 (Week 0): MRI with ASL will be performed either for research alone or along with patient's standard of care imaging session including contrast-enhancement.
  T1 (Day 7+-2): contrast-enhanced research MRI with ASL
Arm/Group | RCC Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Repeatability of Perfusion Measurement in Kidneys
Description: Measurement of perfusion in kidneys in healthy volunteers for the assessment of repeatability.
Time Frame: Baseline, 2 weeks
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 4
ml/100g/min
  Baseline | 306 (60)
  2 weeks | 283 (56)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: This is an observational study, where the participants undergo MR imaging. Hence, the standard time frame for monitoring adverse events is 24 hours.
Arm/Group | RCC Patients | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT04831138/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT04831138/ICF_001.pdf